CLINICAL TRIAL: NCT06228716
Title: The Effect of the Training Given by Hybrid Simulation Method on The Skill and Anxiety Level of the Patients Applying Subcutaneous Biological Drugs
Brief Title: Education With Hybrid Simulation Method in Patients Administering Subcutaneous Biological Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İlayda Türkoğlu (Other)
Responsible Party: Sponsor-Investigator, İlayda Türkoğlu, Msc, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10840098-772.02-E.60612
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Self Administration; Biological Therapy; Training
Keywords: Self administratation; anxiety; subcutaneous injection; biological therapy; simulation training
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research was carried out with a pretest-posttest randomized controlled experimental design to evaluate the effect of the training given by the hybrid simulation method to individuals who self-administer subcutaneous biological drugs on application skills and anxiety levels.
Who Masked: Participant
Masking Description: The individual and the independent observer participating in the subcutaneous biological drug administration skill evaluation were enabled to participate in the evaluation process with a blinding method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subcutaneous biological drug self-administration training was given by the researcher in two stages, theoretical and practical, face to face. Power point presentation and training brochure were used in theoretical training. The practical training given after the theoretical training was given using the Hybrid simulation method. The Wearable Subcutaneous Injection Hybrid Simulator developed by the researcher was worn by the individuals after being informed about its purpose and function. A medicine pen similar to their own medicine pens (demo pen without medicine), dry cotton, alcohol swab (similar to the ones that come in medicine pen boxes), and a small notepad and pen were left in a clean medicine tray on a clean table. Afterwards, they were expected to apply the subcutaneous application step by step as explained to them. Each application step they made incorrectly was corrected and repeated with the support of the researcher.The training took approximately 40 minutes.
  Interventions: Device: Training with hybrid simulation method
- Kontrol Group (Other): Subcutaneous biological drug self-administration training was given theoretically face to face by the researcher using a power point presentation and training brochure. The training lasted approximately 25 minutes and was given in the same room where the experimental group received training.
  Interventions: Other: Broshure

INTERVENTIONS:
Device: Training with hybrid simulation method — Subcutaneous biological drug self-administration training was given by the researcher in two stages, theoretical and practical, face to face. Power point presentation and training brochure were used in theoretical training. The practical training given after the theoretical training was given using the Hybrid simulation method. The Wearable Subcutaneous Injection Hybrid Simulator developed by the researcher was worn by the individuals after being informed about its purpose and function. Afterwards, they were expected to apply the subcutaneous application step by step as explained to them. Each application step they made incorrectly was corrected and repeated with the support of the researcher. The application was considered successful if they completed all application steps correctly from start to finish. The training took approximately 40 minutes. After the practical training, the individuals' questions, if any, were answered and the training was terminated.
  Arms: Experimental
Other: Broshure — Subcutaneous biological drug self-administration training was given theoretically face to face by the researcher using a power point presentation and training brochure. The training lasted approximately 25 minutes and was given in the same room where the experimental group received training. After the training, any questions the individuals had were answered and the training was ended.
  Arms: Kontrol Group

SUMMARY:
In recent years, vital drugs such as heparin, insulin, growth hormone, interferons, monoclonal antibodies and drugs containing proteins that can be destroyed in the gastrointestinal tract have been developed in the form of self-subcutaneous injection in order to reduce the negative effects of treatment practices on the lives of patients. After the training, the patients can apply the subcutaneous injection on their own without assistance. This situation reduces the dependency on the nurse and allows the patient to apply the injection on time, without the need to reach the health institutions. In a study, it is stated that the inadequacy of injection training causes many patients to develop inappropriate injection behavior patterns and to acquire habits regarding these inappropriate techniques. It is also stated that the anxiety they experienced before the injection caused them to ignore the critical steps towards the injection application. In this study, the Subcutaneous Injection Hybrid Model, developed by the researcher, will be used in the training of patients who administer biologic drugs subcutaneously. It is thought that these patients will improve their injection practice skills and reduce their anxiety about injection by repetitive applications by training with the hybrid simulation method.

DETAILED DESCRIPTION:
A poor self-injection experience can lead to undesirable treatment outcomes. However, increasing morbidity and mortality rates are closely related to non-adherence to treatment. Undesirable results due to non-compliance with treatment lead to more visits to emergency services, prolongation of inpatient treatments and increased surgical interventions, thus increasing the workload and costs of health services. In addition, patients who cannot receive repeated and effective training on subcutaneous injection application cause them to experience anxiety about subcutaneous drug administration on their own, and often come to health units only for subcutaneous injection, due to the limited ability to administer. This situation can both negatively affect the daily life activities and self-efficacy perceptions of the patients and increase the workload and cost in health services.

Hybrid Simulation; It is also defined as "patient-centered simulation". In this method; Simulated/standardized patient method is used together with auxiliary tools. Wearable simulation tools are used in this simulation type. When the literature is examined, it is seen that various training methods for self-administration skills are used in patients followed in the rheumatology outpatient clinic, but their effectiveness is controversial. In addition, no study has been found to evaluate the effectiveness of a hybrid simulation-based training on the improvement of application skills and reduction of anxiety regarding subcutaneous injection of biologic drugs, for which adherence to treatment is vital. The aim of this study is to evaluate the effect of training given by simulation method on patients who administer subcutaneous biologic drugs on their application skills and anxiety level. It is thought that these patients, who are trained with the hybrid simulation method, will decrease their negative experiences of subcutaneous biologic drug administration by repetitive applications and incorrect drug administration due to misunderstandings, their injection administration skills will improve, and their anxiety about injection will decrease.

Purpose and Design of the Research

This study was planned in a pre-test-post-test randomized controlled design in order to evaluate the effect of the training given by the hybrid simulation method to the patients who administered subcutaneous biologic drugs on the application skill and anxiety level.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-50,
* Residing in Istanbul,
* Their family/relatives are not using medication in subcutaneous injection form,
* Receiving injection training for the first time,
* First time injection application,
* Using biological medication for the first time,
* Using subcutaneous biological medication for the first time,
* The requested subcutaneous biological drug must be in pen form,
* The drug administration dose should be once every 2 weeks (1/14),
* Being open to communication and cooperation,
* No experience of injecting any living creature (human or animal),
* There is no cognitive, perceptual, or physical disability that would hinder the ability to administer self-injection,
* Volunteering to participate in the research.

Exclusion Criteria:

* Leaving the study at any stage of the research process,
* Not participating in the training and evaluations included in the research,
* Having any local or systemic infectious disease at any stage of the research process.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | Before training
  It was structured by the researcher in line with the literature and included demographic information such as "the individual's name, surname, age, gender, marital status, education level" as well as "medical diagnosis, the name of the subcutaneous medication used and whether he/she has received any simulation-based training before and his phone number." It consisted of 11 questions including ".
Determination of state anxiety level/pretest application | Before training and 2. week before first self administration of subcutaneous injection by the patient
  All individuals in both the experimental and control groups included in the sample were asked to fill out the State Anxiety Scale to evaluate their anxiety levels before the subcutaneous biological drug administration training.
Subcutaneous Biological Drug Self-Administration Skill Checklist | 1. week post training; 2. week post training
  Checklist consisting of 20 application steps to evaluate the skill level of Subcutaneous Biological Drug Self-Administration

SECONDARY OUTCOMES:
Subcutaneous Biological Drug Knowledge Test | 1. week post training
  17-item test assessing the level of knowledge about subcutaneous biological drugs
Patient Education Evaluation Survey | 1. week post training
  5-point Likert-type survey consisting of 10 items on patients' evaluation of education
Trait anxiety scale | 1. week post training
  20-item scale assessing an individual's trait anxiety. trait anxiety scale

CONTACTS AND LOCATIONS:
Overall Officials: İlayda Türkoğlu, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Üsküdar, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenger F, Konig A, Ochsendorf F, Kaufmann R, Pinter A. Correct performance of subcutaneous injections in plaque psoriasis: comparison of trained and untrained patients with different application systems in routine clinical care. J Dermatolog Treat. 2021 Dec;32(8):898-906. doi: 10.1080/09546634.2020.1720580. Epub 2020 Feb 2. PMID 32009495
- [Background] Timmermann H, Mailander C. Home Self-Administration of Biologics - A German Survey among Omalizumab-Treated Patients with Severe Asthma and their Treating Physicians. Pneumologie. 2020 Feb;74(2):103-111. doi: 10.1055/a-1069-0900. Epub 2020 Jan 9. PMID 31935761
- [Result] Fischer-Cartlidge E, Romanoff S, Thom B, Burrows Walters C. Comparing Self-Injection Teaching Strategies for Patients With Breast Cancer and Their Caregivers: A Pilot Study. Clin J Oncol Nurs. 2016 Oct 1;20(5):515-21. doi: 10.1188/16.CJON.515-521. PMID 27668371